CLINICAL TRIAL: NCT01270204
Title: The Effect of Food Taste, Temperature, and Viscosity on Swallowing Efficiency
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 201018116
Record Dates: First submitted 2010-12-16; First posted 2011-01-05 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Dysphagia
Keywords: Dysphagia; Swallowing Problems; Dynamic Fluoroscopic Swallow Study; Aspiration; Regurgitation; Acid Reflux
MeSH Terms: conditions — Deglutition Disorders; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Volunteers: Patients older than 55 years of age with no history of voice, swallowing, reflux, or progressive neurologic disease affecting the swallowing mechanism.
- Patients with Dysphagia: Patients older than 55 years of age with the following condition: Dysphagia (the sensation of swallowing difficulty), globus, gastroesophageal reflux, or any other condition requiring referral for a dynamic swallowing study.

SUMMARY:
The purpose of this study is to evaluate the effect of taste on swallowing efficiency, to evaluate the effect of temperature on swallowing efficiency, and to evaluate the effect of viscosity on swallowing efficiency.

DETAILED DESCRIPTION:
Swallowing problems (dysphagia) are encountered frequently in primary practice and in the hospital setting. The list of possible causes is large, ranging from strokes and neurological disease to complications of cancer treatment, acid reflux, and surgery. Many patients have a reduced ability to feel food and fluid (reduced sensation) within the throat (pharynx) and this leads to an inability to manipulate food and fluids in the correct manner. This can produce a variety of swallowing problems such as choking on foods and fluids, regurgitation, aspiration, weight loss, malnutrition and poor quality of life.

Treatment of dysphagia is largely directed at rehabilitation of muscle power and education about safe swallowing techniques or positioning that limits food and fluid from entering the airway. One of the most widely accepted treatments of dysphagia is to alter the texture of food. Most patients with dysphagia will have more difficulty swallowing thin liquids. By adding a thickener to the liquid, a food bolus becomes more cohesive, and is less likely to become aspirated. Various types of thickening products are available over-the-counter without a prescription. These thickening products are bland and currently have no flavor. We hypothesize that alterations in food taste (sweet, salty, etc…), viscosity, and temperature, will improve swallowing efficiency. The purpose of this investigation is to evaluate the effects of food taste, texture, and temperature on swallowing efficiency. The goal is to develop safer, better tasting food products and improve the quality of life in patients with disabling swallowing disorders.

ELIGIBILITY:
Inclusion Criteria:

* Normal Volunteers:

  * Older than 55 years of age
  * No history of voice, swallowing, reflux, or progressive neurologic disease affecting the swallowing mechanism.
  * A normal self-administered dysphagia questionnaire (EAT-10 score of less than three)
* Patients with Dysphagia

  * Older than 55 years of age
  * Patients with the following condition: Dysphagia, globus, gastroesophageal reflux, or any other condition requiring referral for a dynamic swallowing study.
  * Patients willing to provide written informed consent for their participation in the study.

Exclusion Criteria:

1. Patients unable to complete the administration of the full taste and viscosity protocol.
2. Patients with profound dysphagia unable to safely consume the test solutions.
3. Patients with known sensitivities or allergies to any of the test solutions.
4. Patients who are prisoners.
5. Patients have a history of diabetes.
6. Patients who are unable to follow the simple instructions to swallow the test solutions on instruction and answer the questionnaire.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 dysphagic volunteers and 10 healthy volunteers
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Swallowing amplitude as measured on digital accelerometry. | Measurement is made at the time of patient participation.
  Digital accelerometry is a non-invasive method of measuring swallowing efficiency. A surface sensor is taped to the skin over the region of the thyroid prominence. When the patient swallows, the sensors measures upward acceleration of the thyroid cartilage and a measurement of swallowing amplitude, a surrogate measure for swallowing efficiency, is obtained.

SECONDARY OUTCOMES:
To evaluate swallowing efficiency. | Measurement is taken at the time of patient participation.
  Peak pharyngeal pressure, upper esophageal sphincter (UES) residual pressure, and UES relaxation time, all surrogate measure sof swallowing efficiency, will be measured using pharyngeal manometry.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Belafsky, MD, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Department of Otolaryngology, Sacramento, California, United States